CLINICAL TRIAL: NCT01713166
Title: Effects of Colloid and Crystalloid on the Microcirculatory Alterations During Off-pump Coronary Artery Bypass Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Yunseok Jeon, Associate Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: YSJeon_crystalloid vs colloid
Record Dates: First submitted 2012-10-21; First posted 2012-10-24 (Estimated); Last update posted 2016-06-16 (Estimated); Status verified 2016-06

CONDITIONS: Cardiac Surgery
MeSH Terms: interventions — Hydroxyethyl Starch Derivatives

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Plasmalyte solution (Active Comparator): Plasmalyte solution infusion to meet the fluid requirements.
  Interventions: Drug: plasmalyte solution
- Hextend (Experimental): 6% Hetastarch administeration instead of crystalloids until the total amount given reached 20 ml/kg, which is the maximally allowed daily dose. Afterward, plasmalyte solution infusion to meet the fluid requirements.
  Interventions: Drug: Hextend

INTERVENTIONS:
Drug: plasmalyte solution — plasmalyte solution
  Arms: Plasmalyte solution
Drug: Hextend — Hetastarch administration instead of crystalloids until the total amount given reached 20 ml/kg, which is the maximally allowed daily dose. Afterward, plasmalyte solution infusion to meet the fluid requirements.
  Arms: Hextend

SUMMARY:
The purpose of this study is to compare the effects of crystalloid and colloid, which are used for pump priming solution, on the microcirculatory alterations during cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

* Off-pump Coronary Artery Bypass Surgery

Exclusion Criteria:

* Infection
* Postoperative use of steroid
* Liver cirrhosis, Child-Pugh C
* Renal disease on hemodialysis
* Patients who cannot receive vascular occlusion test (severe peripheral vascular disease, arteriovenous fistula, burn)
* EF < 40% on the preoperative echocardiography
* Preoperative use of vasopressors or inotropic agents

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2013-03; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Recovery slope | until 2 days after surgery
  Recovery slope is a marker of microcirculation. The tissue oxygen saturation (StO2) using InspectraTM StO2 (Hutchinson Technology Inc.,USA) will be recorded continuously. The InspectraTM StO2 probe will be placed on the skin of the thenar eminence and the blood pressure cuff will be wrapped around the arm. After performing vascular occlusion test, the recovery slope will be calculated by the software.
syndecan-1 | until 2 days after surgery
  marker of glycocalyx degradation

SECONDARY OUTCOMES:
lactate | until 2 days after surgery
StO2 (tissue oxygen saturation) | until 2 days after surgery
Cytokine | until 2 days after surgery
  Interleukin (IL)-1b, IL-6, IL-8, IL-10, TNF-a

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea